CLINICAL TRIAL: NCT05118828
Title: Guided Internet-based Interventions in Primary Care: the INTERMENTAL Effectiveness-implementation Randomized Controlled Trial
Brief Title: Guided Internet-based Interventions in Primary Care Effectiveness-implementation Randomized Controlled Trial
Acronym: INTERMENTAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian Directorate of Health (Other Government); University of Bergen (Other); Göteborg University (Other); University of Tromso (Other); Sussex Partnership NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Robert Smith, Research Professor, Norwegian Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-397
Record Dates: First submitted 2021-10-17; First posted 2021-11-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Mild to Moderate Depression
Keywords: Anxiety; Depression; Guided internet-based interventions; CBT; Outcome monitoring; Dissemination; Routine services
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided internet-based treatment (AS-iCBT) (Experimental)
  Interventions: Behavioral: Guided internet-based cognitive behavioural therapy
- Treatment as usual in Prompt Mental Health Care (TAU-PMHC) (Active Comparator)
  Interventions: Behavioral: Treatment as usual in Prompt Mental Health Care (TAU-PMHC)

INTERVENTIONS:
Behavioral: Guided internet-based cognitive behavioural therapy — AS-iCBT offers guided CBT intervention for anxiety and depression, each consisting of 6 modules. It is recommended for clients to complete 1 module weekly. The structure and content of the programme modules follow evidence-based CBT principles, and comprises cognitive and behavioural components such as self-monitoring, gradual stimulus control, exposure, behavioural activation, and cognitive restructuring. It is recommended that therapist support is provided weekly during short sessions that focus on progress monitoring and feedback on completed work. Support sessions should last 15-20 minutes and are preferably delivered by phone or video conference.
  Arms: Guided internet-based treatment (AS-iCBT)
Behavioral: Treatment as usual in Prompt Mental Health Care (TAU-PMHC) — TAU-PMHC includes both low-intensity (guided self-help, group-based psychoeducation) and high-intensity CBT (F2F-CBT). The TAU-PMHC condition basically represents how PMHC services currently operates (i.e. a pragmatic stepped care model) and provides therapists with more flexibility to accommodate client needs and preferences.
  Arms: Treatment as usual in Prompt Mental Health Care (TAU-PMHC)

SUMMARY:
Internet-based cognitive behavioral therapy for anxiety and depression have far-reaching potential to overcome common barriers to accessing evidence-based treatment, such as waiting lists, travel distance and costs. Despite the undeniable promise of iCBT, several aspects remain poorly understood and warrants further study.

The INTERMENTAL project is a joint effort between Norwegian Institute of Public Health, Norwegian Directorate of Health and six Prompt Mental Health Care (PMHC) services, situated in 11 municipalities, to evaluate the iCBT interventions developed by the technology company "Assistert Selvhjelp" (AS-iCBT). We will conduct a large-scale hybrid effectiveness-implementation randomized controlled non-inferiority trial that will provide new knowledge on the effectiveness, cost-effectiveness and implementation of AS-iCBT in primary care.

Primary objective: Examine the non-inferiority of guided internet-based cognitive behavioural treatment "Assistert Selvhjelp" (AS-iCBT) compared to treatment as usual in the primary care service Prompt Mental Health Care (TAU-PMHC) with regard to effects on symptoms of anxiety and depression.

Secondary objectives: (i) Examine the non-inferiority of AS-iCBT compared to TAU-PMHC on other outcomes such as quality of life, functional level, specific anxiety measures (social anxiety, panic disorder), sleep and employment status; (ii) Examine the cost-effectiveness of AS-iCBT compared to TAU-PMHC; (iii) Examine to what extent moderators and mediators of change are associated with treatment effectiveness of AS-iCBT; (iv) Assess whether AS-iCBT is as acceptable and appropriate for treatment of anxiety and depression as TAU-PMHC, and examine barriers/facilitators for their further implementation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anxiety and/or mild to moderate depression.
* Being above 18 years of age and a resident in the pilot sites.
* Basic verbal and oral Norwegian proficiency.
* Having internet access and ability to use it.

Exclusion Criteria:

* Entitled to secondary care services due to eating disorder, suicide risk, bipolar disorder, severe depression, psychotic symptoms, severe substance abuse, and/or personality disorder.
* Two or more previous treatment attempts in secondary care services without effect.
* Serious physical health problem as primary problem.
* Clients that have had treatment at PMHC before and only require a booster session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in mean levels of depression | Baseline to 6-month follow-up
  Changes in mean levels of depression as measured by the Patient Health Questionnaire (PHQ). Scores from 0 to 27, higher scores indicate worse outcome.
Changes in mean levels of anxiety | Baseline to 6-month follow-up
  Changes in mean levels of anxiety as measured by the Generalized Anxiety Disorder scale (GAD). Scores from 0 to 21, higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Changes in mean levels of depression at 12-, 18- and 24-months follow-up | Baseline to 24-month follow-up
  Changes in mean levels of depression as measured by respectively the Patient Health Questionnaire (PHQ). Scores from 0 to 27, higher scores indicate worse outcome.
Changes in mean levels of anxiety at 12-, 18- and 24-months follow-up | Baseline to 24-month follow-up
  Changes in mean levels of anxiety as measured by respectively the Generalized Anxiety Disorder scale (GAD). Scores from 0 to 21, higher scores indicate worse outcome.
Recovery rate at 6-, 12-, 18-, and 24-months follow-up | Baseline to 24-month follow-up
  Proportion of clients that have recovered based on pre-defined cut-offs for PHQ and GAD. Cut-off for PHQ is >= 10 and for GAD >=8.
Work Participation based on questionnaire data | Baseline to 24-month follow-up
  Increased or maintained work participation at 6-, 12-, 18-, and 24-months follow-up, defined as maintained work participation, new employment or a full or partial return-to-work.
Work Participation based on registry data | Baseline to 24-month follow-up
  Increased or maintained work participation at 6-, 12-, 18-, and 24-months follow-up, defined as maintained work participation, new employment or a full or partial return-to-work.
Health-related quality of life | Baseline to 24-month follow-up
  Changes in mean levels of health-related QoL as measured by EuroQol-5D-5L at 6-, 12-, 18-, and 24-months follow-up. Scores from 5 to 25. Higher scores indicate worse outcome.
Mental well-being | Baseline to 24-month follow-up
  Changes in mean levels of mental well-being as measured by the 7-item short Warwick Edinburgh Mental Well-Being Scale (sWEMWBS) at 6-, 12-, 18-, and 24-months follow-up. Scores from 7 to 35. Lower scores indicate worse outcome.
Insomnia | Baseline to 24-month follow-up
  Recovery from insomnia as assessed by a proxy for Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-V) insomnia diagnosis at 6-, 12-, 18-, and 24-months follow-up. The proxy measure is derived from a revised version of the Bergen Insomnia Scale (BIS).
Specific anxiety measure: social anxiety disorder | Baseline to 24-month follow-up
  Changes in mean levels of symptoms of social anxiety disorder as measured by the Social Phobia Inventory (SPIN-9) at 6-, 12-, 18-, and 24-months follow-up. Scores from 9 to 45. Higher scores indicate worse outcome.
Specific anxiety measure: panic disorder | Baseline to 24-month follow-up
  Changes in mean levels of symptoms of panic disorder as measures by the Panic Disorder Screener (PADIS) at 6-, 12-, 18-, and 24-months follow-up. Scores from 0 to 13. Higher scores indicate worse outcome.
Physical activity | Baseline to 24-month follow-up
  Changes in mean levels of physical activity at 6-, 12-, 18-, and 24-months follow-up. Physical activity will be assessed using three sets of questions, assessing the average number of times exercising each week, and the average intensity and average hours each time. This 3-item questionnaire has previously been used in the large population-based Nord-Trøndelag Health Study (the HUNT studies). A physical activity index will be derived in line with the work from Kurtze et al. (2008). Scores from 0 to 15. Lower scores indicate worse outcome.
Sedentary behaviour | Baseline to 24-month follow-up
  Changes in mean levels of sedentary behaviour (SB) at 6-, 12-, 18-, and 24-months follow-up. Sedentary behaviour was assessed using two questions assessing the average number of hours of sedentary behaviour during the last two weeks. The first questions covers sedentary behaviour during weekdays, whereas the second question covers sedentary behaviour during the weekend. A weighted sum score of these items is used to derive an index for SB. The items are based on the single item on SB in the short form of the international physical activity questionnaire (IPAQ-SF). Scores from 0 to 5. Higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smith, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (6):
- Norway (6):
  - PMHC Fosen, Brekstad
  - PMHC Karmøy, Kopervik
  - PMHC Vestvågøy, Leknes
  - PMHC Notodden, Notodden
  - PMHC Sandnes, Sandnes
  - PMHC Modum, Vikersund

IPD SHARING:
Plan to Share IPD: No